CLINICAL TRIAL: NCT01561391
Title: An Open-Label, Randomized, Parallel, Multicenter Trial Comparing the Safety and Efficacy of rFVIIa When Administered as i.v. Bolus or i.v. Continuous Infusion to Hemophiliacs With Inhibitors During and After Major Surgery
Brief Title: Safety and Efficacy of Activated Recombinant Human Factor VII in Haemophilia Patients With Inhibitors During and After Major Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F7HAEM/USA/4/USA
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor IX; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous infusion (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Bolus injection (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Control (Experimental)
  Interventions: Other: factor IX; Drug: factor VIII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Infused continuously at 50 mcg/kg/hr through Day 5 then at 25 mcg/kg/hr on Days 6 to10.
  Arms: Continuous infusion
Drug: activated recombinant human factor VII — Injected every 2 hours during surgery through Day 5, then every 4 hours for Days 6 to 10.
  Arms: Bolus injection
Other: factor IX — Patients with haemophilia A or B without inhibitors undergoing similar surgery were treated in accordance with local standard of care per physician's orders.
  Arms: Control
Drug: factor VIII — Patients with haemophilia A or B without inhibitors undergoing similar surgery were treated in accordance with local standard of care per physician's orders.
  Arms: Control

SUMMARY:
This trial is conducted in North America. The aim of this trial is to compare the safety and efficacy of activated recombinant human factor VII in patients with haemophilia A or B undergoing major surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Have haemophilia A or B with inhibitors to factor VIII or IX, respectively
* Have had a historical inhibitor level of at least five Bethesda units or have had an inadequate haemostatic response to 250 U/kg of factor VIII or IX or have had an inadequate response to FEIBA
* Require pre-planned major surgery in hospital

Exclusion Criteria:

* Have participated in or have been treated with any investigational drug other than activated recombinant human factor VII within the last thirty days
* Have been treated with any haemostatic agent, including rFVIIa, within 48 hours of preoperative dose
* Have any haemostatic disorder other than haemophilia

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1998-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Presence and maintenance of haemostasis
Changes in FVII:C (Factor VII clotting activity) levels following administration of activated recombinant human factor VII

SECONDARY OUTCOMES:
Adverse Events
Changes in coagulation-related parameters

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- United States (12):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Rochester, Minnesota
  - Novo Nordisk Investigational Site, New Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas

REFERENCES:
- [Result] Pruthi RK, Mathew P, Valentino LA, Sumner MJ, Seremetis S, Hoots WK; NovoSeven in Surgery Study Investigators. Haemostatic efficacy and safety of bolus and continuous infusion of recombinant factor VIIa are comparable in haemophilia patients with inhibitors undergoing major surgery. Results from an open-label, randomized, multicenter trial. Thromb Haemost. 2007 Oct;98(4):726-32. PMID 17938794
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com